CLINICAL TRIAL: NCT00944788
Title: Feasibility and Impact on Quality of Life and Depressive Symptoms of a Structured Qi-gong Program for Hospitalized Older Adults. A Pilot Study.
Brief Title: A Structured Qi-gong Program for Hospitalized Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacio Salut i Envelliment UAB (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: FICE09071; CEEAH_UAB_792H
Record Dates: First submitted 2009-07-22; First posted 2009-07-23 (Estimated); Last update posted 2013-06-13 (Estimated); Status verified 2013-06

CONDITIONS: Quality of Life; Behavioral Symptoms; Patient Compliance
Keywords: physical activity; aging; inpatients; quality of life; depression
MeSH Terms: conditions — Behavioral Symptoms; Patient Compliance; Motor Activity; Depression | interventions — Qigong

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- qi-gong (Experimental)
  Interventions: Other: qi-gong
- Usual care (No Intervention)

INTERVENTIONS:
Other: qi-gong — Physical activity similar to tai-chi
  Arms: qi-gong

SUMMARY:
The purpose of this study is to test the effects on a number of health outcomes and the feasibility of a structured program of qi-gong, a form of tai-chi which has been previously tested in older populations, in older hospitalized patients. In particular, this pilot study aims to assess changes in quality of life and depressive symptoms after 4 weeks of treatment, with the hypothesis that this intervention will have a positive impact on these two domains, compared to usual care. Adherence will be also monitored in the intervention arm.

ELIGIBILITY:
Inclusion Criteria:

* >=50 years old
* Preserved ability to move inside the house (also using walking aids or chair)
* Estimation of at least one month of hospitalization (convalescence or rehabilitation)
* Ability and willing to sign informed consent

Exclusion Criteria:

* Moderate to severe cognitive impairment (SPMSQ >= 4)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2009-07; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Quality of life | 4 weeks

SECONDARY OUTCOMES:
Depressive symptoms | 4 weeks
Adherence | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Marco Inzitari, MD, PhD, Principal Investigator — Fundació Institut Català de l'Envelliment
Locations (1):
- Parc Sanitari Pere Virgili, Barcelona, Spain

REFERENCES:
- [Background] Rogers CE, Larkey LK, Keller C. A review of clinical trials of tai chi and qigong in older adults. West J Nurs Res. 2009 Mar;31(2):245-79. doi: 10.1177/0193945908327529. PMID 19179544
- [Derived] Martinez N, Martorell C, Espinosa L, Marasigan V, Domenech S, Inzitari M. Impact of Qigong on quality of life, pain and depressive symptoms in older adults admitted to an intermediate care rehabilitation unit: a randomized controlled trial. Aging Clin Exp Res. 2015 Apr;27(2):125-30. doi: 10.1007/s40520-014-0250-y. Epub 2014 Jun 14. PMID 24927783